CLINICAL TRIAL: NCT07220668
Title: Sense4Safety Intervention
Acronym: Sense4Safety
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GM1XX56LEP58; 1R01AG090377-01A1 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment
Keywords: fall prevention; mild cognitive impairment; exercise training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants receive no interventional component, standard care
- Intervention Group (Experimental): Participants receive the Sense4Safety Intervention
  Interventions: Behavioral: Sense4Safety

INTERVENTIONS:
Behavioral: Sense4Safety — Sense4Safety is a technology-enhanced intervention that includes multiple components: 1) in-home assessment; 2) tailored education and exercise; 3) passive monitoring and communication. The intervention is primarily via video-conferencing or phone, supplemented by in-home visits at intake, and 6 months to conduct in-person assessments.
  Other Names: Fall Prevention Intervention
  Arms: Intervention Group

SUMMARY:
Falls and fall-related injuries are significant public health issues for adults 65 years of age and older. Over a third of older adults (OA) fall each year and 10-20% of falls result in serious injuries such as fractures and head trauma. The annual direct medical costs in the US as a result of falls are estimated to exceed $50 billion, and this estimate does not include the indirect costs of disability, dependence, and decreased quality of life. This project targets community dwelling OA with mild cognitive impairment (MCI). MCI is a leading risk factor for falls in OA. Approximately 15%-20% of OA have MCI, and over 60% of OA with MCI fall annually - two to three times the rate of those without cognitive impairment. We have developed and pilot-tested an innovative technology-supported intervention called Sense4Safety to 1) identify escalating risk for falls real-time through in-home passive sensor monitoring; 2) employ machine learning to inform individualized alerts for fall risk; and 3) link 'at risk' older adults with a coach who will guide them in implementing evidence-based individualized plans to reduce fall-risk. The purpose of this study is to assess the effectiveness of Sense4Safety in reducing fall risk with a randomized clinical trial, and understand implementation factors to improve the scalability of Sense4Safety in diverse community settings.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* reside in senior living communities and plan to be in the area for more than 6 months
* be able to walk household distances
* score of at least 1 of 12 on the Short Physical Performance Battery (SPPB)
* meet MCI criteria (MCI is defined as a score ≥17 Montreal Cognitive Assessment)

Exclusion Criteria:

Exclusion criteria include terminal illness, central nervous system condition such as stroke or Parkinson's disease, diagnosis of dementia, severe vision or hearing deficits, and reliant on wheelchair or scooter within living quarters.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | 0, 3 and 6 months
  Usual gait speed (m/s)
Lower extremity strength and functional mobility | 0, 3, 6 mos.
  Instrumented 30-second chair stand
Functional mobility and fall risk | 0, 3, 6 mos.
  Instrumented Timed Up & Go (TUG) Test
Static balance in narrow stance positions | 0, 3, 6 mos.
  Instrumented 90-second balance test

SECONDARY OUTCOMES:
Fear of Falling | 0, 3, 6 mos.
  measures the level of concern about falling during 16 social and physical activities inside and outside the home whether or not the person actually does the activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No